CLINICAL TRIAL: NCT02990468
Title: A Phase 1 / Phase 2 Trial of Concurrent Radiation Therapy, Cisplatin, and BMX-001 in Locally Advanced Head and Neck Cancer
Brief Title: A Trial of Concurrent Radiation Therapy, Cisplatin, and BMX-001 in Locally Advanced Head and Neck Cancer
Acronym: BMX-HN
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioMimetix JV, LLC (Industry)
Collaborators: Duke University (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BMX-HN-001
Record Dates: First submitted 2016-11-28; First posted 2016-12-13 (Estimated); Results first posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-02

CONDITIONS: Head and Neck Cancer
Keywords: Mucositis; Xerostomia
MeSH Terms: conditions — Head and Neck Neoplasms; Mucositis; Xerostomia | interventions — Radiotherapy; Cisplatin

STUDY DESIGN:
Intervention Model Description: Dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Radiation Therapy, Cisplatin and BMX-001 (Experimental): In Phase 1, safety and tolerability of BMX-001 will be assessed using a Continual Reassessment Method and a maximum tolerated dose (MTD) will be determined using a single arm design. In Phase 2, the severity of radiation-induced mucositis and xerostomia will be assessed using a single arm design.
  Interventions: Drug: BMX-001; Radiation: Radiation Therapy; Drug: Cisplatin

INTERVENTIONS:
Drug: BMX-001 — Subcutaneous injection.
Radiation: Radiation Therapy — Patients will receive standard dose intensity modulated radiation therapy (IMRT).
Drug: Cisplatin — Cisplatin will be administered per institution's standard of care practice.

SUMMARY:
This is a Phase 1 / Phase 2 study of newly diagnosed patients with biopsy-proven head and neck cancer (squamous cell carcinoma) who are undergoing standard radiation therapy and treatment with cisplatin. BMX-001 added to radiation therapy and cisplatin is expected to reduce radiation-induced mucositis and xerostomia and also has the potential to benefit the survival of head and neck cancer patients. In Phase 1, safety and tolerability of BMX-001 will be assessed using a Continual Reassessment Method (CRM) and a maximum tolerated dose (MTD) will be determined. BMX-001 will be given subcutaneously first with a loading dose zero to four days prior to the start of chemoradiation and followed by twice a week doses at one-half of the loading dose for the duration of radiation therapy plus two weeks. In Phase 2 both safety and efficacy of BMX-001 will be evaluated. Impact on mucositis and xerostomia will also be assessed. A maximum of 48 patients will be enrolled to the MTD dose determined in Phase 1 to confirm the MTD. The investigators hypothesize that BMX-001 when added to standard radiation therapy and cisplatin will be safe at pharmacologically relevant doses in patients with newly diagnosed head and neck cancer. The investigators also hypothesize that in Phase 2 of this study the addition of BMX-001 will reduce the severity of radiation-induced mucositis and xerostomia in patients receiving head and neck radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed diagnosis of squamous cell carcinoma of the oropharynx, larynx, hypopharynx, or oral cavity with clinical or pathologic high-risk features for whom cisplatin and radiation would be considered appropriate care.
2. Treatment plan to receive a continuous course of IMRT delivered as single daily fractions of 2.0 to 2.1 Gy with a cumulative radiation dose between 60 Gy and 70 Gy depending on whether patients are considered post-operative high risk or unresectable/organ preservation high risk. Planned radiation treatment fields must include at least two oral sites buccal mucosa, retromolar trigone, floor of mouth, oral tongue, soft palate, hard palate) with a portion of each site receiving a minimum total of 50 Gy.
3. Patients who are to undergo definitive chemoradiation must have clinically or radiographically evident measurable disease at the primary site and/or at nodal stations. Tonsillectomy or local excision of the primary without removal of nodal disease is permitted.
4. Limited neck dissections retrieving ≤ 4 nodes are permitted and considered as non-therapeutic nodal excisions. Fine needle aspirations of the neck that are positive for squamous cell carcinoma are sufficient for diagnosis pending pathology review at participating institutions.
5. For patients undergoing curative intent resection the following criteria are required:

   * Pathologically (histologically or cytologically) proven diagnosis of head and neck squamous cell carcinoma
   * Patients must have undergone gross total surgical resection within 42 days prior to registration and beginning of therapy under the clinical trial. Note: Patients may have biopsy under general anesthesia in an operating room followed by definitive ablative cancer surgery representing gross total resection.
6. Clinical or pathologic stage Stage III-IVb per the American Joint Committee on Cancer (AJCC), 7th edition.
7. General history and physical examination by a radiation oncologist and medical oncologist within 4 weeks prior to enrollment.
8. Examination by an ear/nose/throat (ENT) or head and neck surgeon, including laryngopharyngoscopy (mirror and/or fiberoptic and/or direct procedure) within 8 weeks prior to enrollment.
9. Zubrod Performance Status 0-2 within 4 weeks prior to enrollment
10. Complete blood count (CBC)/differential obtained within 7 days prior to starting the study drug with adequate bone marrow function, defined as follows:

    * Hemoglobin ≥ 9.0 g/dl;
    * Platelets ≥ 100,000 cells/mm3;
    * Absolute neutrophil count (ANC) > 1,500 cell/mm3.
11. Adequate hepatic function as defined as follows:

    * Total bilirubin < 2x institutional upper limit of normal (ULN) within 7 days prior to starting the study drug;
    * Aspartate aminotransferase (AST) and AST <3x institutional ULN within 7 days prior to starting the study drug.
12. Adequate renal function defined as follows:

    * Serum creatinine < 1.5 mg/dl within 7 days prior to starting the study drug or creatinine clearance rate (CCr) ≥ 50 mL/min within 7 days prior to starting the study drug determined by 24-hour collection or estimated by Cockcroft-Gault formula:

    CCr male = [(140 - age) x (wt in kg)]/[(Serum Cr mg/dl) x (72)] CCr female = 0.85 x (CrCl male)
13. Negative pregnancy test for women of child-bearing potential within 48 hours prior to first dose of BMX-001.
14. Women of childbearing potential and male participants must agree to use a medically effective means of birth control throughout their participation in the treatment phase of the study and until 12 months following the last study treatment.

Exclusion Criteria:

1. Stage I or II; T1N1 and T2N1 stage III presentations per AJCC 7th edition
2. Distant metastasis
3. Hypertension requiring 3 or more anti-hypertensive medications to control
4. Grade ≥2 hypotension at screening
5. Requirement for concurrent treatment with nitrates or other drugs that may, in the judgment of the treating investigator, create a risk for a precipitous decrease in blood pressure
6. History of syncope within the last 6 months
7. Patients receiving, or unable to stop use at least 1 week prior to receiving the first dose of BMX-001, medications listed in Section 12.2 of the protocol are not eligible.
8. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic
9. Women who are breast feeding are not eligible
10. Prior allergic reaction to cisplatin
11. Known hypersensitivity to compounds of similar chemical composition to BMX-001
12. Grade 3-4 electrolyte abnormalities (CTCAE v 4.03) except sodium, which must be ≥126 mmol/L.
13. Prior unrelated malignancy requiring current active treatment with the exception of cervical carcinoma in situ, basal cell carcinoma of the skin, resected T1-2N0M0 differentiated thyroid cancers, invasive cancers with a 3-year disease-free interval, Ta bladder cancers, or low and favorable intermediate risk prostate cancer.
14. Prior history of HNSCC receiving radiation or chemo-radiation.
15. Prior systemic chemotherapy for the study cancer (including neoadjuvant chemotherapy); note that prior chemotherapy for a different cancer is allowable.
16. Prior radiotherapy that would result in overlap of radiation treatment fields with planned treatment for study cancer.
17. Severe, active co-morbidity, defined as follows:

    * Cardiovascular disease or cerebrovascular disease, for example cerebrovascular accidents or myocardial infarction ≤ 6 months prior to study enrollment, unstable angina, New York Heart Association (NYHA) Grade II or greater congestive heart failure (CHF), or serious cardiac arrhythmia uncontrolled by medication or with the potential to interfere with protocol treatment;
    * Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months prior to enrollment;
    * History or evidence upon physical/neurological examination of central nervous system disease (e.g., seizures) unrelated to cancer unless adequately controlled by medication;
    * Acute bacterial or fungal infection requiring intravenous antibiotics within 7 days of enrollment;
    * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days of registration;
    * Patients known to be HIV positive or have active viral hepatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of California San Francisco, San Francisco, California
  - University of Florida- Gainesville, Gainesville, Florida
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: Group 1: Participants were administered a 7 mg loading dose followed by a 3.5 mg maintenance dose twice a week for up to 8 weeks while receiving concurrent cisplatin and RT.
- Phase 1: Group II: Participants were administered a 14 mg loading dose followed by a 7 mg maintenance dose twice a week for up to 8 weeks while receiving concurrent cisplatin and RT.
- Phase 2: Group III - MTD: Participants were administered a 28 mg loading dose followed by a 14 mg maintenance dose twice a week for up to 8 weeks while receiving concurrent cisplatin and RT.
Period: Phase 1: Dose Escalation
Arm/Group | Phase 1: Group 1 | Phase 1: Group II | Phase 2: Group III - MTD
Started | 3 | 3 | 0
Completed | 3 | 3 | 0
Not Completed | 0 | 0 | 0
Period: Phase 2: MTD
Arm/Group | Phase 1: Group 1 | Phase 1: Group II | Phase 2: Group III - MTD
Started | 0 | 0 | 23
Completed | 0 | 0 | 22
Not Completed | 0 | 0 | 1
Not completed — Change in treatment | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: dose escalation
Groups:
- Phase 1: Group I: Subjects were administered a 7 mg loading dose subcutaneously followed by a 3.5 mg maintenance dose subcutaneously twice a week while on concurrent cisplatin and RT.
- Phase 1: Group II: Subjects were administered a 14 mg loading dose subcutaneously followed by a 7 mg maintenance dose subcutaneously twice a week while on concurrent cisplatin and RT.
- Phase 2: Group III: Subjects were administered a 28 mg loading dose subcutaneously followed by a 14 mg maintenance dose subcutaneously twice a week while on concurrent cisplatin and RT.
- Total: Total of all reporting groups
Arm/Group | Phase 1: Group I | Phase 1: Group II | Phase 2: Group III | Total
Number analyzed (Participants) | 3 | 3 | 23 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 15 | 17
  >=65 years | 2 | 2 | 8 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.33 (12.97) | 67.67 (4.91) | 60.96 (7.66) | 61.28 (8.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 3 | 4
  Male | 2 | 3 | 20 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 3 | 23 | 29
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 23 | 29

OUTCOME MEASURES:

1. Primary Outcome: Assess the Safety of the Study Drug by Calculating the Proportion of Patients Who Experience Grade 4 or 5 Study Drug Related Adverse Events, as Assessed by CTCAE v 4.03.
Description: This outcome is to confirm the safety and tolerability of escalating doses of BMX-001 in conjunction with RT and concurrent cisplatin in a cohort of newly diagnosed patients with locally advanced head and neck cancers. Each dose will be reported separately.
Time Frame: 1 year
Population: Each dosing group reported seperately.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1: Group 1: Subjects were administered a 7 mg loading dose subcutaneously followed by a 3.5 mg maintenance dose subcutaneously twice a week while on concurrent cisplatin and RT.
Arm/Group | Phase 1: Group 1 | Phase 1: Group II | Phase 2: Group III
Number analyzed (Participants) | 3 | 3 | 23
Participants | 0 | 0 | 0

2. Primary Outcome: Incidence Radiation-induced Mucositis by Clinician Scoring
Description: Mucositis will be scored using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. Higher scores are indicative of worse symptoms. Grade 0-5. We are reporting the incidence of the patients that had mucositis grade 1-5.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Group 1 | Phase 1: Group II | Phase 2: Group III
Number analyzed (Participants) | 3 | 3 | 23
Participants | 1 | 1 | 10

3. Secondary Outcome: Incidence of Radiation-induced Xerostomia by Stimulated Saliva Production
Description: Xerostomia will also be assessed by measurement of stimulated saliva production posttreatment.
Time Frame: 6 months
Population: one subject in group 3 did not complete follow up and was excluded from analysis
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Phase 1: Group 1 | Phase 1: Group II | Phase 2: Group III
Number analyzed (Participants) | 3 | 3 | 22
gram | 1.487 (0.144) | 2.387 (0.688) | 2.115 (1.151)

4. Secondary Outcome: Incidence of Radiation-induced Xerostomia by Unstimulated Saliva Production
Description: Xerostomia will also be assessed by measurement of unstimulated saliva production post treatment.
Time Frame: 6 months
Population: one subject in group 3 did not complete follow up and was excluded from analysis
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Phase 1: Group 1 | Phase 1: Group II | Phase 2: Group III
Number analyzed (Participants) | 2 | 2 | 22
gram | 0.42 (0.041) | 1.090 (0.334) | 1.255 (0.932)

5. Secondary Outcome: Incidence of Radiation-induced Xerostomia by Clinician Scoring
Description: Xerostomia will be assessed using Maximum Xerostomia Clinical Score Common Terminology Criteria for Adverse Events (CTCAE) 4.03. Scores range from 0 to 5 with 0 being no xerostomia and 5 being the worst. Mean maximum xerostomia grade of patients assessed is reported.
Time Frame: 6 months
Population: One subject in group 3 did not complete follow up and was excluded from the analysis (a score of 0 representing no xerostomia)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Phase 1: Group 1 | Phase 1: Group II | Phase 2: Group III
Number analyzed (Participants) | 3 | 3 | 22
score on a scale | 1 (0) | 1.33 (0.27) | 1.29 (0.13)

6. Secondary Outcome: Duration of Radiation-induced Mucositis
Description: Mucositis will be scored using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. Duration of Oral Mucositis WHO Grade 3 or higher measured as the days of severe oral mucositis.
Time Frame: 6 month 6 months
Population: only the patients that had mucositis were evaluated for duration
Measure: Mean (Standard Error); unit: days
Arm/Group | Phase 1: Group 1 | Phase 1: Group II | Phase 2: Group III
Number analyzed (Participants) | 1 | 1 | 10
days | 22 (NA) — The sample size is too small to calculate standard error. | 18 (NA) — The sample size is too small to calculate standard error. | 37.4 (8.2)

7. Secondary Outcome: To Examine the Impact on Radiation Dermatitis When Adding BMX-001 to Treatment
Description: To examine the impact on radiation dermatitis of BMX-001 in combination with RT and concurrent cisplatin at 30-39 Gy, 40-49 Gy, 50-59 Gy, and 60-70 Gy, the duration of radiation dermatitis, and evaluation of radiation dermatitis-related patient-reported outcomes
Time Frame: 30 days
Population: Data was not collected or analyzed
Arm/Group | Phase 1: Group 1 | Phase 1: Group II | Phase 2: Group III
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the time the subject signs the informed consent form through and of treatment visit (one year follow up)
Description: An AE can therefore be any unfavorable and unintended or worsening sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of BMX-001, whether or not related to use of the BMX-001. Abnormal laboratory findings without clinical significance (based on the PI's judgment) should not be recorded as AEs, but laboratory value changes that require therapy or adjustment in prior therapy are considered adverse events.
Arm/Group | Phase 1: Group I | Phase 1: Group II | Phase 2: Group III
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 11/23
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Group I (N=3) | Phase 1: Group II (N=3) | Phase 2: Group III (N=23)
Abdominal Infection (Gastrointestinal disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1
Febrile neutropenia (Renal and urinary disorders) | 0 | 0 | 1
Gastronomy failure (Gastrointestinal disorders) | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Lung infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Neutropenic colitis (Gastrointestinal disorders) | 0 | 0 | 1
Presyncope (Vascular disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 3
Sepsis (Infections and infestations) | 1 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Group I (N=3) | Phase 1: Group II (N=3) | Phase 2: Group III (N=23)
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 3
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 4
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 15
Anal incontinence (Gastrointestinal disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 5
Blood creatinine increased (Investigations) | 0 | 0 | 5
Candida infection (Infections and infestations) | 0 | 0 | 3
Chills (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4
Conduction Disorder (Cardiac disorders) | 1 | 0 | 0
Confusional State (Nervous system disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 3 | 19
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Deafness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 6
Dehydration (Metabolism and nutrition disorders) | 3 | 3 | 13
Depression (Psychiatric disorders) | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2
Dizziness (Nervous system disorders) | 1 | 1 | 10
Dry eye (Eye disorders) | 0 | 1 | 0
Dry Mouth (Gastrointestinal disorders) | 3 | 3 | 20
Dysgeusia (Nervous system disorders) | 3 | 3 | 20
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 7
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 13
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 6
Early satiety (Gastrointestinal disorders) | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 5
Fatigue (General disorders) | 3 | 3 | 21
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Feeling jittery (General disorders) | 0 | 0 | 2
Flushing (Vascular disorders) | 0 | 0 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 3 | 16
Hypertension (Vascular disorders) | 0 | 0 | 2
Hypoacusis (Ear and labyrinth disorders) | 1 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 2
Hypoalbuminaemia (Hepatobiliary disorders) | 0 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 9
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 6
Hypotension (Vascular disorders) | 0 | 0 | 3
Hypothyroidism (Endocrine disorders) | 1 | 0 | 2
Influenza like illness (General disorders) | 0 | 0 | 3
Infusion site extravasation (General disorders) | 0 | 0 | 2
Injection site bruising (General disorders) | 0 | 0 | 3
Injection site reaction (General disorders) | 3 | 3 | 19
Insomnia (Nervous system disorders) | 0 | 1 | 3
Lip infection (Infections and infestations) | 1 | 0 | 2
Lip pain (Gastrointestinal disorders) | 0 | 1 | 0
Localised oedema (General disorders) | 1 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 2
Lymphoedema (Blood and lymphatic system disorders) | 1 | 2 | 11
Malaise (General disorders) | 1 | 0 | 0
Middle ear adhesions (Ear and labyrinth disorders) | 0 | 1 | 0
Mucosal infection (Infections and infestations) | 2 | 2 | 9
Mucosal inflammation (General disorders) | 0 | 0 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 3 | 3 | 19
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 4
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 3
Neutrophil count decreased (Investigations) | 0 | 1 | 12
Non-cardiac chest pain (General disorders) | 0 | 0 | 2
Odynophagia (Gastrointestinal disorders) | 0 | 2 | 11
Oedema (General disorders) | 0 | 0 | 3
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 2
Oral pain (Gastrointestinal disorders) | 0 | 0 | 5
Oropharyngeal pain (Gastrointestinal disorders) | 3 | 2 | 15
Otitis externa (Ear and labyrinth disorders) | 0 | 1 | 0
Pain (General disorders) | 2 | 1 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 3 | 0
Platelet count decreased (Investigations) | 0 | 2 | 17
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 9
Pyrexia (General disorders) | 1 | 1 | 3
Radiation skin injury (Injury, poisoning and procedural complications) | 3 | 3 | 16
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Salivary duct inflammation (Gastrointestinal disorders) | 3 | 3 | 13
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 8
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Skin infection (Infections and infestations) | 1 | 0 | 2
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 3 | 3 | 15
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 2 | 8
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 3 | 7
Weight decreased (Investigations) | 2 | 1 | 17
White blood cell count decreased (Investigations) | 0 | 0 | 17

LIMITATIONS AND CAVEATS:
This was a dose escalation study with all subjects receiving the intervention. There was no control arm for comparison. This will be addressed in a future clinical trial. This study design was effective for a safety, dose-escalation study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/68/NCT02990468/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/68/NCT02990468/ICF_001.pdf